CLINICAL TRIAL: NCT00346346
Title: Longitudinal Analysis of the B-Cell Immune Response to Plasmodium Falciparum in Mali
Brief Title: Analysis of the Immune Response to the Malaria Parasite in Mali, West Africa
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906147; 06-I-N147
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2013-01-23

CONDITIONS: Malaria
Keywords: Immunity; Memory; ELISPOT; Malaria; Prospective
MeSH Terms: conditions — Malaria

SUMMARY:
This study will examine the immune response to the malaria parasite at the cellular level to better understand why people achieve natural immunity to the parasite only after multiple infections and why immunity diminishes rapidly in the absence of ongoing infection. The results of this study may provide insight into whether and how natural immunity can be improved upon by vaccination.

Healthy people 2-4 and 18-25 years of age who live in the village of Kambila, Mali, may be eligible for this 1-year study. Participants have a small blood sample collected from a vein in the arm and also from two finger pricks at the beginning of the study, then every 2 months for 6 months and at the end of the study (for a total of five samples). People who become ill with malaria are evaluated and treated by a physician. Those recovering from their first episode of malaria during the study period have another blood sample collection and two finger pricks (bringing to six the total number of samples collected).

DETAILED DESCRIPTION:
Malaria remains an important public health threat, responsible for over one million deaths annually, the majority among African children. The development of a safe and effective vaccine is widely regarded as a crucial step forward in the control of this disease. However, vaccines tested in clinical trials to date have resulted in very short-lived protection at best. This appears to mirror the kinetics of naturally acquired immunity to Plasmodium falciparum, in that multiple infections are required over many years before clinical immunity is achieved, and then appears to diminish relatively rapidly in the absence of ongoing infection. The mechanisms underlying the delayed acquisition and presumably rapid loss of humoral immunity are poorly understood. A more detailed understanding of these processes on the cellular level may provide insight into whether and how natural immunity can be improved upon by vaccination. This longitudinal cohort study in a P. falciparum endemic village of Mali proposes to test the hypothesis that resistance to malaria is associated with acquisition of P. falciparum specific memory B cells. The 52 week study will cover an entire malaria transmission season and will enroll 224 healthy persons ages 2 to 10 and 18 to 25. After informed consent is obtained from the participant, or the participant's parent or guardian, an age appropriate volume of venous blood will be drawn at baseline, and at 2, 4, 6, and 12 months thereafter; and serum and peripheral blood mononuclear cells (PBMC) will be frozen and stored. One convalescent blood sample per participant will also be drawn within two weeks of their first symptomatic P. falciparum infection. Clinical data, including the frequency and severity of malaria infections, will be collected during the study period by passive surveillance. After 52 weeks, serum and PBMC will be thawed and analyzed to determine antibody titers to malaria antigens and to enumerate relevant B cell subpopulations, including total and antigen-specific naive, memory, and plasma cells by ELISPOT assays and flow cytometry.

ELIGIBILITY:
* INCLUSION CRITERIA - HEALTHY VOLUNTEERS AT ENROLLMENT:

  1. Males and females ages 2 to 10 years or 18 to 25 years.
  2. Will be living in Kambila for one year and available for 12 month follow-up.
  3. Willing to have blood specimens stored.
  4. Willingness of adult volunteer to participate in the study as evidenced by the completed informed consent document.
  5. Willingness of parent or guardian to have his or her child participate in the study as evidenced by the completed informed consent document.

EXCLUSION CRITERIA - HEALTHY VOLUNTEERS AT ENROLLMENT:

1. Active bleeding or hematocrit less than or equal to 15 % (for both children and adults).
2. Fever greater than 38 degrees C, or systemic illness at enrollment.
3. Currently using anti-malarial medications.
4. The following two exclusion items may not have occurred in the last 30 days: participation in a vaccine or drug trial, or use of corticosteroid or other immunosuppressive drugs.
5. Current pregnancy or a plan to become pregnant during the one year study period. Pregnancy status will be determined at enrollment by urine dipstick, and at subsequent time points by self-report only.
6. While on this protocol, if a subject enrolls in another study that requires the administration of experimental therapies (vaccines or medications), he/she may no longer participate in this protocol.

(Presence of P. falciparum parasitemia in the absence of symptoms at the time of screening is not exclusionary).

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 237 (Actual)
Dates: Start 2006-04-17; Study Completion 2013-01-23

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Crompton, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Achidi EA, Perlmann H, Salimonu LS, Perlmann P, Walker O, Asuzu MC. A longitudinal study of seroreactivities to Plasmodium falciparum antigens in Nigerian infants during their first year of life. Acta Trop. 1995 May;59(2):173-83. doi: 10.1016/0001-706x(95)00076-q. PMID 7676908
- [Background] ALLISON AC. Protection afforded by sickle-cell trait against subtertian malareal infection. Br Med J. 1954 Feb 6;1(4857):290-4. doi: 10.1136/bmj.1.4857.290. No abstract available. PMID 13115700
- [Background] ALLISON AC. Glucose-6-phosphate dehydrogenase deficiency in red blood cells of East Africans. Nature. 1960 May 14;186:531-2. doi: 10.1038/186531a0. No abstract available. PMID 13792821